CLINICAL TRIAL: NCT01110265
Title: Attention Training and Its Effects on Body Image Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Evelyn Smith, The University of Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USydney11760
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Body Dissatisfaction; Eating Disorder Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo training (Placebo Comparator)
  Interventions: Behavioral: placebo training
- attention training (Experimental)
  Interventions: Behavioral: attention training

INTERVENTIONS:
Behavioral: attention training
  Arms: attention training
Behavioral: placebo training
  Arms: placebo training

SUMMARY:
Research has consistently found attentional biases towards negative weight-related stimuli in individuals with eating disorders. It has been suggested that these biases may act as a vulnerability factor for the development and maintenance of body dissatisfaction and may therefore be an important target for intervention. Previous studies have demonstrated the capacity to modify the patterns of attention allocation to threatening stimuli in a variety of anxiety disorders, with a subsequent and sustained reduction in anxiety symptoms. Thus, the present study aimed at testing the efficacy of attention training in reducing attentional biases and eating disorder symptoms in individuals with elevated levels of body image disturbance and eating disorder symptomatology of clinical severity. Thirty-two participants were randomly allocated to receive eight sessions of a 10-minute computer task aimed at training their attention away from weight-related stimuli or a control placebo training condition. Results showed that participants in the attention training group had a significantly greater reduction in their attentional bias and body dissatisfaction from pre- to post-training relative to the placebo condition. At follow-up, both groups showed a significant decrease in body dissatisfaction from their pre-training levels. The only significant difference between groups in eating disorder symptoms at follow-up was in terms of the attention training group experiencing a greater reduction in weight and shape concerns.

ELIGIBILITY:
Inclusion Criteria:

* If they have a score on the Body Shape Questionnaire of 113 or more AND a score in the EDE-Q of 4 or more in any subscale.

Exclusion Criteria:

* attention bias score of <-10

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Sydney, Sydney, New South Wales, Australia